CLINICAL TRIAL: NCT04657510
Title: Femoral frACturEs and COVID-19. Retrospective Comparative Cohort Study on the Early Prognosis of Patients Affected by Proximal Femur Fractures and COVID-19.
Brief Title: Femoral frACturEs and COVID-19.
Acronym: FACE COVID-19
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio (Other)
Responsible Party: Sponsor
Other Study IDs: FACE COVID-19
Record Dates: First submitted 2020-11-14; First posted 2020-12-08 (Actual); Last update posted 2020-12-08 (Actual); Status verified 2020-12

CONDITIONS: Covid19; Femur Fracture; Fragility Fracture
Keywords: proximal femur fracture; fragility fracture; Covid-19; SARS-CoV2; FACE-COVID 19; prognosis; cohort study
MeSH Terms: conditions — COVID-19; Femoral Fractures; Proximal Femoral Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Proximal femur fracture AND COVID-19: Surgical treatment of femur fracture
  Interventions: Other: COVID-19
- Proximal femur fracture NO COVID: Surgical treatment of femur fracture
  Interventions: Other: COVID-19

INTERVENTIONS:
Other: COVID-19 — Patients affected versus not affected by COVID-19, with the same starting condition (proximal femur fracture)

SUMMARY:
Retrospective cohort study comparing the early prognosis after surgically-treated proximal femur fragility fractures in patients affected and not affected by COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥45 years
* Admitted to IRCCS Orthopaedic Institute Galeazzi for proximal femur fractures from march 2020 to april 2020.
* Tested for COVID-19 through naso-pharyngeal swab analized with RT-PCR

Exclusion Criteria:

* Age <45 years
* Not tested for SARS-CoV-2
* Other fractures (including bilateral proximal femur fractures)

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with >45 years of age admitted to our center from march 2020 to april 2020 for proximal femur fracture and tested for SARS-CoV-2.
Sampling Method: Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2020-11-14 (Actual); Primary Completion 2020-12-01 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Survival at discharge day (comparison between the two groups) | on discharge day, on average after 1 week
  Survival at discharge day (comparison between the two groups)

SECONDARY OUTCOMES:
Length of stay (comparison between the two groups) | on discharge day, on average 1 week
  Length of stay (comparison between the two groups)
Readmission rate (comparison between the two groups) | up to 30 days after discharge
  Readmission rate (comparison between the two groups)
Complications rate (comparison between the two groups) | up to 30 days after discharge
  Complications rate (comparison between the two groups)
Survival at 30 days after discharge (comparison between the two groups) | 30 days after discharge
  Survival at 30 days after discharge (comparison between the two groups)
Routine lab exams values (comparison between the two groups) | At admission, 1st postoperative day, 5th postoperative day, on discharge day
  Routine lab exams values (comparison between the two groups)

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe M Peretti, MD, Principal Investigator — IRCCS Istituto Ortopedico Galeazzi
Locations (1):
- IRCCS Istituto Ortopedico Galeazzi, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided